CLINICAL TRIAL: NCT04865822
Title: Single Session Pain Education for Chronic Pain
Brief Title: Single Session Pain Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Heather Poupore-King, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 59054
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Education (Experimental): Participant will attend a single session pain education course
  Interventions: Behavioral: Single session pain education class
- wait list control (No Intervention): Participants will be wait listed then receive intervention

INTERVENTIONS:
Behavioral: Single session pain education class — Pain education classes will be provided in person group or virtual settings
  Arms: Pain Education

SUMMARY:
To pilot single session pain education classes aimed at improving outcomes and behaviors in patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain patients, pain longer than 3 months
* ability to adhere to and complete study protocols

Exclusion Criteria:

* not fluent in English
* recent injury at the discretion of the researcher
* previous completion of pain education class at the discretion of the researcher
* current cancer diagnosis or other medical condition at the discretion of the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in Tampa scale for kinesiophobia at three months | month 3
  TSK is a measure of kinesiophobia in people who have chronic pain

IPD SHARING:
Plan to Share IPD: No